CLINICAL TRIAL: NCT01593592
Title: Lactobacillus Reuteri in Management of Helicobacter Pylori Infection in Dyspeptic Patients: a Double Blind Placebo Controlled Randomized Clinical Trial
Brief Title: Lactobacillus Reuteri in Management of Helicobacter Pylori Infection in Dyspeptic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Moahmed Hassan Emara, Lecturer of Tropical Medicine and Hepatogastroenterology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#:395/29-4-2012; IRB#:395/29-4-2012 (Other: Zagazig University)
Record Dates: First submitted 2012-05-05; First posted 2012-05-08 (Estimated); Results first posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-07

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Lactobacillus reuteri; dyspeptic patients; eradication
MeSH Terms: interventions — Omeprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus reuteri group (Experimental): The active group that will receive the standard triple therapy and Lactobacillus reuteri
  Interventions: Dietary Supplement: Lactobacillus reuteri; Drug: Omeprazole; Drug: Amoxicillin; Drug: Clarithromycin
- Control group (Placebo Comparator): The control group that will receive the standard triple therapy and placebo
  Interventions: Dietary Supplement: Placebo; Drug: Omeprazole; Drug: Amoxicillin; Drug: Clarithromycin

INTERVENTIONS:
Dietary Supplement: Lactobacillus reuteri — Will receive triple therapy (omeprazole 20 mg b.i.d., amoxicillin 1000 mg b.i.d, clarithromycin 500mg b.i.d) and L. reuteri (is a mixture of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475, will be delivered a dose of 1x108 CFU each strain, means giving daily chewable tablet containing 2x108 CFU/day) for 2 weeks followed by L. reuteri for another 2 weeks.
  Arms: Lactobacillus reuteri group
Dietary Supplement: Placebo — Will receive triple therapy (omeprazole 20 mg b.i.d., amoxicillin 1000 mg b.i.d, clarithromycin 500mg b.i.d) and a placebo (1.5 mg per dose as chewable tablets) for 2 weeks followed by placebo for another 2 weeks.
  Arms: Control group
Drug: Omeprazole — All patients will receive omeprazole 20 mg b.i.d for 2 week
Drug: Amoxicillin — amoxicillin 1000 mg b.i.d for 2 weeks
Drug: Clarithromycin — clarithromycin 500mg b.i.d for 2 weeks

SUMMARY:
Addition of L. reuteri to the standard triple therapy improves H. Pylori treatment outcomes.

DETAILED DESCRIPTION:
Helicobacter pylori (H. Pylori) infection is a wide spread disease and is endemic in many countries including Egypt with a wide range of morbidity; that requires appropriate antimicrobial therapy . However, worldwide the eradication rate following the standard triple therapy is declining and this may necessitates introduction of new antimicrobial agents . On the sight of bearing in vivo and in vitro activity against H. Pylori, the use of different strains of probiotics in treatment of H. Pylori may be thus justifiable, Lactobacillus reuteri (L. reuteri) which through different mechanisms including production of reuterin have anti H.pylori activity have been tried in improving the eradication rates of H.pylori with contradictory results . This study is conducted to test the assumption that addition of L. reuteri to the standard triple therapy in treatment of H. Pylori improves the eradication rates and clinical aspects in H. Pylori infection.

ELIGIBILITY:
Inclusion Criteria:

Inclusion of patients with these criteria

1. Age: 18-60 years
2. Any sex
3. Confirmed H. Pylori infection defined by pathological lesions and either histopathological confirmation of the organism, rapid urease test or H. Pylori antigen in stool
4. Good mentality to understand aim, benefits and steps of the study
5. Assumed availability during the study period
6. Written informed consent

Exclusion Criteria:

* Exclusion of

  1. Patients with chronic diseases e.g. diabetes, renal failure, cirrhosis…etc.
  2. Patients with malignancy.
  3. Patients with gall bladder disorders.
  4. Patients with peptic ulcer.
  5. Patients with prior upper GIT surgery.
  6. Patients with probiotics therapy in the last one month.
  7. Patients with triple therapy, antibiotics, proton pump inhibitors and H2 receptor blockers therapy within one month.
  8. Patients with known allergy to the used medications

     -

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqia Province, Egypt

REFERENCES:
- See also: Study location Hospital — http://www.hosp.zu.edu.eg/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All adult dyspeptic patients presented to outpatient gastroenterology clinics of the Tropical Medicine and Internal Medicine Departments, Faculty of Medicine, Zagazig University Hospitals, Egypt from June 2012 to February 2013 were offered to share in the study
Groups:
- Control Group: The control group that will receive the standard triple therapy and placebo
  Placebo : Will receive triple therapy (omeprazole 20 mg b.i.d., amoxicillin 1000 mg b.i.d, clarithromycin 500mg b.i.d) and a placebo (1.5 mg per dose as chewable tablets) for 2 weeks followed by placebo for another 2 weeks.
- Lactobacillus Reuteri Group: The active group that will receive the standard triple therapy and Lactobacillus reuteri
  Lactobacillus reuteri : Will receive triple therapy (omeprazole 20 mg b.i.d., amoxicillin 1000 mg b.i.d, clarithromycin 500mg b.i.d) and L. reuteri (is a mixture of L. reuteri DSM 17938 and L. reuteri ATCC PTA 6475, will be delivered a dose of 1x108 CFU each strain, means giving daily chewable tablet containing 2x108 CFU/day) for 2 weeks followed by L. reuteri for another 2 weeks.
Period: Overall Study
Arm/Group | Control Group | Lactobacillus Reuteri Group
Started | 35 | 35
Completed | 35 | 35
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All were dyspeptic patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus Reuteri Group | Control Group | Total
Number analyzed (Participants) | 35 | 35 | 70
Age, Continuous [Mean (Full Range); unit: years] | 33.20 [18 to 60] | 36.80 [22 to 60] | 35.00 [18 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 24 | 46
  Male | 13 | 11 | 24
ِAge [Mean (Standard Deviation); unit: years] — It is a measure of age from 18 to 60 years old for participants
  years | 33.20 (13.974) | 36.80 (11.085) | 35.00 (12.650)

OUTCOME MEASURES:

1. Primary Outcome: Eradication of H Pylori Infection 4 Weeks After Completion of Therapy
Description: H. pylori eradication is defined in this study as concomitant negativity to all previously positive tests (H. pylori antigen in stool; histopathological confirmation of H. pylori bacilli; and rapid urease test.) 4 weeks after the end of therapy.
Time Frame: 4 weeks therapy
Population: It is assessment of all the 70 participants about H pylori eradication status
Measure: Number; unit: participants
Arm/Group | Control Group | Lactobacillus Reuteri Group
Number analyzed (Participants) | 35 | 35
participants | 23 | 26

2. Secondary Outcome: Severe Adverse Effects to the Used Medications and Dietary Supplements.
Time Frame: 4 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Control Group | Lactobacillus Reuteri Group
Number analyzed (Participants) | 35 | 35
percentage of participants | 0 | 0
Statistical Analysis 1: Comparison: Control Group vs Lactobacillus Reuteri Group; A total of 70 patients were included; 35 in each arm. The sample size was calculated assuming eradication of H. pylori in at least 70% of treated patients, aiming to detect a difference of 30% based on a 0.80 power to detect significant difference (p =0.05, two-sided); Test type: Superiority or Other; percentage = 0

3. Secondary Outcome: The Secondary End Point Was the Development of Severe Adverse Effects to the Used Medications and Dietary Supplements.
Description: Severe adverse effects to the used medications and dietary supplements, these may expose the participants to major morbidity and may change the outcomes in them.
Time Frame: 8 weeks
Measure: Number; unit: participants
Arm/Group | Control Group | Lactobacillus Reuteri Group
Number analyzed (Participants) | 35 | 35
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: Patients were followed up for 8 weeks to report any adverse events and side effects
Arm/Group | Lactobacillus Reuteri Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35
Other Adverse Events (participants affected / at risk) | 10/35 | 25/35
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lactobacillus Reuteri Group (N=35) | Control Group (N=35)
Galactorrhea (Reproductive system and breast disorders) | 0 | 1 — one virgin female patient developed galactorrhea
Taste disorders (Gastrointestinal disorders) | 2 | 8
Diarrhea (Gastrointestinal disorders) | 1 | 10
Distension (Gastrointestinal disorders) | 5 | 4
Vomiting (Gastrointestinal disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
no limitations

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No